CLINICAL TRIAL: NCT01949428
Title: A Field Study to Observe Symptom Scores and Allergy Medication Usage in Subjects With a History of House Dust Mite-Induced Rhinoconjunctivitis
Brief Title: House Dust Mite Observational Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Pharm-Olam International (Industry)
Responsible Party: Sponsor
Other Study IDs: TH003
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Rhinoconjunctivitis
Keywords: HDM Allergy; Rhinoconjunctivitis

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HDM-Induced Rhinoconjunctivitis Subjects

SUMMARY:
A Field Study to Observe Symptom Scores and Allergy Medication Usage in Subjects with a History of House Dust Mite-Induced Rhinoconjunctivitis

DETAILED DESCRIPTION:
House Dust Mites (HDM) are arachnids that infest bedding, carpet, upholstered furniture and fabric. Like many other allergens, exposure to HDMA in sensitised patients is associated with poorer lung function, greater medication requirements and more asthma symptoms as well as chronic rhinosinusitis symptoms. In contrast to other allergens, there is evidence that HDMA leads to the development of asthma, in addition to exacerbating pre-existing asthma in HDM-sensitised patients.

The proposed observational study is designed to gather information on subjects with HDM-related rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years
* A history of moderate to severe rhinoconjunctivitis (sneezing, rhinorrhoea, itchy nose, nasal blockage, and/or itchy/watery/red/sore eyes) consistent with allergy to HDM for at least 1 year.
* Non-asthmatic, or asthma controlled by Step 1 or 2 treatment as defined by GINA for at least one month.
* Subjects must have a 7-day reflective TRSS (i.e., reflective over the previous 7 days) of ≥12 and must have a score of ≥2 in at least two of the individual symptom components.
* Subjects must have Der p or Der f specific IgE ≥0.35 kU/L as measured by ImmunoCAP®. A blood draw for HDM-specific IgE must be performed during the Screening period.
* Subjects must have Der p or Der f specific IgE ≥0.35 kU/L as measured by ImmunoCAP®. A blood draw for HDM-specific IgE must be performed during the Screening period.

Exclusion Criteria:

* Clinically significant confounding symptoms of allergy to relevant local seasonal allergens (e.g., ragweed, mugwort, tree, grass, mountain cedar, mould) and cannot complete the Screening and Observation period outside the respective allergy seasons.
* Previous immunotherapy treatment with any HDMA for more than 1 month within 5 years prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a History of House Dust Mite-Induced Rhinoconjunctivitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To Document the combined Total Rhinocnjunctivitis Systom Scores (TRSS) and Total allergy medication score | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pharm-Olam, Mississauga, Ontario, Canada